CLINICAL TRIAL: NCT03094260
Title: Interest of Light Therapy in the Treatment of Binge Eating Disorder: Prospective Controlled Randomized Double-blind Trial
Brief Title: Light Therapy and Binge Eating Disorder Treatment (BED Light Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 69HCL16_0626; 2016-A01768-43 (Other: ID-RCB)
Record Dates: First submitted 2017-03-09; First posted 2017-03-29 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Binge-Eating Disorder
MeSH Terms: conditions — Binge-Eating Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High intensity light therapy (Experimental): Treatment with light therapy in high intensity (10,000 lux)
  Interventions: Device: High intensity bright light therapy
- Low intensity light therapy (Placebo Comparator): Treatment with light therapy in low intensity (<500 lux)
  Interventions: Device: Low intensity light therapy

INTERVENTIONS:
Device: High intensity bright light therapy — Treatment with light therapy in high intensity (10,000 lux), daily for 30 days between 6 am and 9 am for 30 minutes.
  Le device is placed at arm's length (at approximately 50-75cm from the eyes) within the field of vision. The light must bathe the face To ensure the light reaches your eyes, this appliance has a stand that can be set to a variable angle. If subject is sitting higher or standing and the top edge of the appliance is below eye level, the appliance will be placed in a tilted position so that its light points further upwards and reaches the eyes. If subject is sitting at a table or desk and the top edge of the appliance is above eye level. The appliance can be placed in a more upright position.
  Arms: High intensity light therapy
Device: Low intensity light therapy — Treatment with light therapy in low intensity (<500 lux), daily for 30 days between 6 am and 9 am for 30 minutes.
  Le device is placed at arm's length (at approximately 50-75cm from the eyes) within the field of vision. The light must bathe the face To ensure the light reaches your eyes, this appliance has a stand that can be set to a variable angle. If subjectis sitting higher or standing and the top edge of the appliance is below eye level, the appliance will be placed in a tilted position so that its light points further upwards and reaches the eyes. If subject is sitting at a table or desk and the top edge of the appliance is above eye level. The appliance can be placed in a more upright position.
  Arms: Low intensity light therapy

SUMMARY:
Binge Eating Disorder (BED) is the most widespread food behavior disorder, with prevalence three times higher than anorexia. Its pathophysiology remains poorly understood and the investigators have few therapeutic options. Following a review of the literature, the investigators hypothesize that luminotherapy could be an innovative treatment of BED by its favorable effect on triggers of hyperphagic access, circadian disturbances, attention and impulsivity. The study is prospective, interventional, randomized, double-blind, monocentric (HCL). 52 patients with BED will be randomized to an active arm with intensive luminotherapy (1 daily 30 min, 10,000 lux in the morning) versus a placebo arm (<500 lux). Treatment will be delver every day during 30 days. Assessments will take place on D0, D30 and D60. The main objective is to compare the evolution of the number of hyperphagic access before and after treatment between the two groups. Secondary objectives are to compare characteristics of hyperphagic access, bodily concerns, food dependence and impulsivity, mood, anxiety, cognitive and attentional profiles (STROOP, Go / No Go, SST, BART, Prospective Time Estimation Task, Switching Task), liking / wanted for different food categories and carbohydrate metabolism (CRP, glucose, insulinemia, insulin resistance, profile of lipid abnormalities, 25-OH vitamin D3).

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 55 years old
* Binge eating disorders or other eating disorders according to DSM V criteria
* Patient with BES score (with " Bing Eating Scale " ) > 18
* Patient with BMI > 18.5 kg/m2
* Patient who agrees to be included in the study and who signs the informed consent form
* Patient affiliated to a healthcare insurance plan

Exclusion Criteria:

* Patients with other psychiatric comorbidities, including a disorder bipolar mood
* Unstabilized diabetic patient with or retinopathy
* Patient with sleep disorder (delay or phase inversion)
* Patient with psychotropic treatment unstabilized (except anxiolytic treatment)
* Recent eye surgery or eye problem preventing exposure to bright light.
* Medication making the skin more sensitive to light (eg. Tablets against malaria)
* Patient who does not understand French/is unable to give consent
* Mentally unbalanced patients, under supervision or guardianship
* Patient already included in a research study
* Pregnancy or desire to be pregnant during the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2018-03-29 (Actual); Primary Completion 2020-04-09 (Actual); Study Completion 2020-04-09 (Actual)

PRIMARY OUTCOMES:
Comparison of the number of hyperphagic access, over 7 consecutive days, before starting therapy with light therapy and discontinuation of treatment | Day-7 to Day-1 period (before Day 0) compared to Day23 to Day30 period (after Day 0)
  The number of hyperphagic access will be determined using a crisis agenda filled out by patients each day

SECONDARY OUTCOMES:
Comparison of the number of hyperphagic access, over 7 consecutive days, before starting therapy with light therapy and 30 days after discontinuation of treatment | Day-7 to Day-1 period compared to Day23 to Day30 period
  The number of hyperphagic access will be determined using a crisis agenda filled out by patients each day
Characteristics of hyperphagic access (severity of the disorder) | Day 0
  Evaluation of the severity of bulimic hyperphagia by the Bing Eating Scale.
Characteristics of hyperphagic access (severity of the disorder) | Day 30
  Evaluation of the severity of bulimic hyperphagia by the Bing Eating Scale.
Characteristics of hyperphagic access (severity of the disorder) | Day 60
  Evaluation of the severity of bulimic hyperphagia by the Bing Eating Scale.
Characteristics of hyperphagic access (duration of crisis) | Day 0
  Evaluation of the duration,by the crisis agenda.
Characteristics of hyperphagic access (duration of crisis) | Day 30
  Evaluation of the duration,by the crisis agenda.
Characteristics of hyperphagic access (duration of crisis) | Day 60
  Evaluation of the duration,by the crisis agenda.
Characteristics of hyperphagic access (amount of food ingested ) | Day 0
  Evaluation of the quantity of food ingested during the hyperphagic access and the delays between two accesses by the crisis agenda.
Characteristics of hyperphagic access (amount of food ingested ) | Day 30
  Evaluation of the quantity of food ingested during the hyperphagic access and the delays between two accesses by the crisis agenda.
Characteristics of hyperphagic access (amount of food ingested ) | Day 60
  Evaluation of the quantity of food ingested during the hyperphagic access and the delays between two accesses by the crisis agenda.
Characteristics of hyperphagic access ( evolution of factors triggering) | Day 0
  Evaluation of the factors triggering by the "START" scale.
Characteristics of hyperphagic access ( evolution of factors triggering) | Day 30
  Evaluation of the factors triggering by the "START" scale.
Characteristics of hyperphagic access ( evolution of factors triggering) | Day 60
  Evaluation of the factors triggering by the "START" scale.
Characteristics of hyperphagic access (severity of the disorder, duration of crisis, amount of food ingested and evolution of factors triggering) | Day 30
  Evaluation of the severity of bulimic hyperphagia by the Bing Eating Scale. Evaluation of the duration, the quantity of food ingested during the hyperphagic access and the delays between two accesses by the crisis agenda. Evaluation of the factors triggering by the "START" scale.
Comparison of the number of hyperphagic access, over 7 consecutive days, before starting therapy with light therapy and 30 days after discontinuation of treatment | Day-7 to Day-1 period (before Day 0) compared to Day53 to Day60 period (after Day 0)
  The number of hyperphagic access will be determined using a crisis agenda filled out by patients each day
Symptomatic development of BED | Day 0
  The symptomatic development of BED will be measured by evaluating :
  * The psychopathology of the BED from the Eating Disorder Inventory 2 questionnaire
  * The Body concerns based on the "Body sharpe" questionnaire
  * The Addiction to food from the Yale Food Addiction scale
  * The Diet-related impulsivity from the Three-Factor Eating Questionnaire
Symptomatic development of BED | Day 30
  The symptomatic development of BED will be measured by evaluating the composite:
  * The psychopathology of the BED from the Eating Disorder Inventory 2 questionnaire
  * The Body concerns based on the "Body sharpe" questionnaire
  * The Addiction to food from the Yale Food Addiction scale
  * The Diet-related impulsivity from the Three-Factor Eating Questionnaire
Symptomatic development of BED | Day 60
  The symptomatic development of BED will be measured by evaluating the composite:
  * The psychopathology of the BED from the Eating Disorder Inventory 2 questionnaire
  * The Body concerns based on the "Body sharpe" questionnaire
  * The Addiction to food from the Yale Food Addiction scale
  * The Diet-related impulsivity from the Three-Factor Eating Questionnaire
Evolution of other psychological parameters related to BED | Day 0
  The evolution of other psychological parameters will be measured by evaluating the composite :the mood from the Beck Depression Inventory scale, the anxiety from the "State Trait Anxiety Inventory or STAI-Y" scale, the clinical impulsivity from the "UPPS-P shortcut" scale
Evolution of other psychological parameters related to BED | Day 30
  The evolution of other psychological parameters will be measured by evaluating the composite the mood from the Beck Depression Inventory scale, the anxiety from the "State Trait Anxiety Inventory or STAI-Y" scale, the clinical impulsivity from the "UPPS-P shortcut" scale
Evolution of other psychological parameters related to BED | Day 60
  The evolution of other psychological parameters will be measured by evaluating the composite mood from the Beck Depression Inventory scale, the anxiety from the "State Trait Anxiety Inventory or STAI-Y" scale, the clinical impulsivity from the "UPPS-P shortcut" scale
Evolution of attentional cognitive profiles and impulsivity | Day 0
  The evolution of attentional and impulsive cognitive profiles will be measured from a computerized neurocognitive test battery whose order will be randomly fixed. The tests will be STROOP, The Go / No Go, The Stop Signal Task, The Balloon Analog Risk Task, The Prospective Time Estimation Task, The Set Switching Task
Evolution of attentional cognitive profiles and impulsivity | Day 30
  The evolution of attentional and impulsive cognitive profiles will be measured from a computerized neurocognitive test battery whose order will be randomly fixed. The tests will be STROOP, The Go / No Go, The Stop Signal Task, The Balloon Analog Risk Task, The Prospective Time Estimation Task, The Set Switching Task
Evolution of attentional cognitive profiles and impulsivity | Day 60
  The evolution of attentional and impulsive cognitive profiles will be measured from a computerized neurocognitive test battery whose order will be randomly fixed. The tests will be STROOP, The Go / No Go, The Stop Signal Task, The Balloon Analog Risk Task, The Prospective Time Estimation Task, The Set Switching Task
Evolution of appetite for different categories of food | Day 0
  The evolution of appetite for different categories of food will be measured from a computerized task: the Leed Food Preference Questionnaire (LFPQ). A description of the test is available at: https://www.millisecond.com/download/library/
Evolution of appetite for different categories of food | Day 30
  The evolution of appetite for different categories of food will be measured from a computerized task: the Leed Food Preference Questionnaire (LFPQ). A description of the test is available at: https://www.millisecond.com/download/library/
Evolution of appetite for different categories of food | Day 60
  The evolution of appetite for different categories of food will be measured from a computerized task: the Leed Food Preference Questionnaire (LFPQ). A description of the test is available at: https://www.millisecond.com/download/library/
Biological parameters may be impacted or mediated by part of the treatment efficiency | Day 0
  Inflammation parameters, glucose, insulinemia, insulin resistance, Profile of lipid abnormalities, 1-25-OH vitamin D3
Biological parameters may be impacted or mediated by part of the treatment efficiency | Day 30
  Inflammation parameters, glucose, insulinemia, insulin resistance, Profile of lipid abnormalities, 1-25-OH vitamin D3
Weight (kilogramm) | Day 0
  Weight will be expressed in absolute value
Weight (kilogramm) | Day 30
  Weight will be expressed in absolute value
Weight (kilogramm) | Day 60
  Weight will be expressed in absolute value
Observance rate to light therapy | day1 to day30
  The assessment of the adherence rate will be quantified by the average number of lux received over the 30 days of treatment. The exposure (expressed in lux number / session) in lux will be measured and recorded using a luxmeter

CONTACTS AND LOCATIONS:
Overall Officials: Diane MORFIN, MD, Principal Investigator — Hospices Civils de Lyon Centre REférent pour l'Anorexie et les Troubles du Comportement Alimentaire de Lyon (CREATyon)
Locations (1):
- HCL Centre REférent pour l'Anorexie et les Troubles du Comportement Alimentaire de Lyon (CREATyon), Bron, France

IPD SHARING:
Plan to Share IPD: No